CLINICAL TRIAL: NCT03922828
Title: Lung Nodule Prospective Database
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/2596
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Lung Neoplasms; Lung Cancer; Lung Adenocarcinoma
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT scans — CT surveillance, Lung biopsy, Lung resection

SUMMARY:
Lung cancer is one of the most common cancers in the Singapore population, being the 2nd most commonly diagnosed cancer amongst males and 3rd most commonly diagnosed cancer amongst females. Pulmonologists, oncologists and thoracic surgeons are often consulted for the evaluation of imaging-identified pulmonary nodules. These may have been identified either incidentally or through screening. The majority of these are indeterminate and definitive investigation with biopsy or resection is invasive and not without risk. Hence, current consensus guidelines adopt a largely expectant strategy in the management of these indeterminate pulmonary nodules.

There is substantial evidence that lung cancer in Asians may be unique with multiple driver mutations, lower age of presentation and may be independent of tobacco exposure. In addition, there are guidelines that recommend that the management of lung nodules in Asia should account for these differences. However, the evidence for alternative recommendations is lacking.

The aim of the study will be to identify radiological and clinical predictors that can improve the diagnosis of lung nodules. These predictors may help build a model for lung nodule evaluation and surveillance.

Prospective database of subjects meeting all of the following inclusion criteria to participate in this study.

1. Evidence of lung nodule on chest radiograph or Computed Tomography regardless of underlying aetiology
2. Age ³ 21 years old
3. Ability to provide informed consent This study will collect existing or prospective data that is part of standard clinical care from the electronic medical record of patients (ambulatory and inpatient from May 2018-2023.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE

   Lung cancer is one of the most common cancers in the Singapore population, being the 2nd most commonly diagnosed cancer amongst males and 3rd most commonly diagnosed cancer amongst females. Pulmonologists, oncologists and thoracic surgeons are often consulted for the evaluation of imaging-identified pulmonary nodules. These may have been identified either incidentally or through screening. The majority of these are indeterminate and definitive investigation with biopsy or resection is invasive and not without risk. Hence, current consensus guidelines adopt a largely expectant strategy in the management of these indeterminate pulmonary nodules.

   There is substantial evidence that lung cancer in Asians may be unique with multiple driver mutations, lower age of presentation and may be independent of tobacco exposure. In addition, there are guidelines that recommend that the management of lung nodules in Asia should account for these differences. However, the evidence for alternative recommendations is lacking.
2. HYPOTHESIS AND OBJECTIVES

   The aim of the study will be to identify radiological and clinical predictors that can improve the diagnosis of lung nodules. These predictors may help build a model for lung nodule evaluation and surveillance.
3. EXPECTED RISKS AND BENEFITS

   There are likely to be no benefits to subjects. They will not be subject to any novel therapy and their clinical/radiological data will only be collected.

   Risks are minimal because patients are subject to only standard diagnostic work-up and existing clinical data collected. There will be no new additional interventions, consultations or hospital visits. They will be asked to complete validated quality of life surveys that will be included into the clinical record.
4. STUDY POPULATION

   4.1. List the number and nature of subjects to be enrolled.

   Patients will only be enrolled from those who present to Singapore General Hospital, National Cancer Centre, National Heart Centre, Changi General Hospital and Sengkang General Hospital (either in an ambulatory or inpatient setting). There is no exclusion of women or minorities. Children are excluded because lung nodule detection in them is rare and the pathological processes, as well as clinical considerations are different.

   4.2. Criteria for Recruitment and Recruitment Process

   Subjects will be recruited if they already have radiographic evidence of a lung nodule.

   4.3. Inclusion Criteria

   The subject must meet all of the following inclusion criteria to participate in this study.
   1. Evidence of lung nodule on chest radiograph or Computed Tomography regardless of underlying aetiology
   2. Age > 21 years old
   3. Ability to provide informed consent

   4.4. Exclusion Criteria Subjects who no radiographic evidence of lung nodules or who are unwilling/unable to provide informed consent
5. STUDY DESIGN AND PROCEDURES/METHODOLOGY

   This study will collect existing or prospective data that is part of standard clinical care
   * Source of the data: electronic medical record of patients (ambulatory and inpatient)
   * Data will be collected prospectively.
   * Time period: May 2018-2023
   * When subject collection is complete, the data will be de-identified and kept in an electronic database
   * Only principal investigator and co-investigators will have access to collected information.
   * Data be kept for 6 years after completion of study for data analysis and manuscript preparation
   * All electronic copies of data will be destroyed at the end of the study. All manual records if any will be shredded.

   Data that will be collected
   * Demographic data such as age, gender, ethnicity, ambulatory/inpatient setting
   * Clinical data including co-morbidities, medication history, American Society of Anaesthesiologists (ASA) status, smoking history, functional status (eg ECOG),
   * Risk factors such as BMI, exercise intensity, previous malignancy, radiation exposure, 2nd hand cigarette exposure, Family history of cancer, asbestos/environmental exposure
   * Radiographic data including nodule size, location and characteristics (borders, density, calcification, cavitation thickness), fibrosis, adenopathy
   * Laboratory data including LDH, glucose, albumin, total protein; Full blood counts, Renal panel, Liver Panel, Coagulation studies
   * Histopathology and microbiology results
   * Procedure details: designation of operator, procedure duration, anaesthesia used, complications, number of biopsies taken, size of specimen, location of procedure, use of anti-microbials

   Subjects may withdraw voluntarily from participation in the study at any time. They will have standard care as indicated by the managing physician
6. SAFETY MEASUREMENTS 6.1. Definitions

   An adverse event (AE) is any untoward medical occurrence that occurs as a result of the study. This will reported to CRIB.

   6.2. Collecting, Recording and Reporting of Adverse Events and Serious Adverse Events to CIRB

   PI will be responsible for submitting to the approving CIRB the completed serious AE Reporting Form within 7 calendar days after the investigator is aware of the event, followed by a complete report within 8 additional calendar days. AE that are related events should be reported at least annually (together with Study Status Report for annual review).

   6.3. Safety Monitoring Plan

   Not applicable. Current standard investigations and treatment to be provided to all subjects.

   6.4. Complaint Handling

   Complaints about the study will be escalated to the clinical Head of Department and included in reports to the CIRB.
7. DATA ANALYSIS

   7.1. Data Quality Assurance

   Data collection will be done by the investigators through the clinical team managing the patient to ensure completion and accuracy.

   7.2. Data Entry and Storage
   * Data will be entered and stored in a secure web application (REDCap)/password controlled hospital computer. When subject data collection is complete, the data will be de-identified and kept in an electronic database (password secured) for analysis. Only investigators will have access to the data.
   * There are no plans to keep any documentation of patients beyond the informed consent forms. These will be stored in the locked department office of the investigators.
8. SAMPLE SIZE AND STATISTICAL METHODS

   8.1. Determination of Sample Size

   The sample size is determined by the number of patients accrued into the database during the study period. As this is a non-comparative study, study size calculation not applicable.

   8.2. Statistical and Analytical Plans
   * Continuous safety analyses tracking for AE
   * Interim Analyses of data on an annual basis
9. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

   The CRIB will be permitted to audit the database as needed. Source documents are from electronic medical records.
10. QUALITY CONTROL AND QUALITY ASSURANCE

    Data collection will be done by the investigators through the clinical team managing the patient to ensure completion and accuracy.
11. ETHICAL CONSIDERATIONS

    11.1. Informed Consent

    Informed consent will be sought from the patient or legal guardian (in the case of minors) by the study investigators before any data collection is done.

    11.2. Confidentiality of Data and Patient Records
    * Data will be entered and stored in a secure web application (REDCap)/password controlled hospital computer. When subject data collection is complete, the data will be de-identified and kept in an electronic database (password secured) for analysis. Only investigators will have access to the data.
    * There are no plans to keep any documentation of patients beyond the informed consent forms. These will be stored in the locked department office of the investigators.
12. PUBLICATIONS

    Investigators will be involved in authorship depending on the degree of contribution.
13. RETENTION OF STUDY DOCUMENTS

    Study documents will be retained for 6 years after the end of the study in a locked department office and hospital computer that is password protected.
14. FUNDING and INSURANCE

This study has no funding.

ELIGIBILITY:
Inclusion Criteria:

* The subject must meet all of the following inclusion criteria to participate in this study.

  1. Evidence of lung nodule on chest radiograph or Computed Tomography regardless of underlying aetiology
  2. Age > 21 years old
  3. Ability to provide informed consent

Exclusion Criteria:

* Subjects who no radiographic evidence of lung nodules or who are unwilling/unable to provide informed consent

Ages: 21 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with lung nodules
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Histology | 3 years
  Malignant or benign

CONTACTS AND LOCATIONS:
Locations (1):
- Singhealth Institutions, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plan to share individual patient data